CLINICAL TRIAL: NCT01428219
Title: A Phase II Trial of Cabozantinib (XL184) in Patients With Castrate-Resistant Prostate Cancer Metastatic to Bone
Brief Title: Trial of Cabozantinib (XL184) in Castrate-Resistant Prostate Cancer Metastatic to Bone
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to slowing enrollment and negative results of a phase III trial using cabozantinib.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2011.069; HUM00052320 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2011-08-30; First posted 2011-09-02 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer Metastatic
Keywords: Prostate; Cancer; Metastatic
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabozantinib (XL184) (Experimental): Cabozantinib is available in capsule form. The dose is 60 mg daily by mouth. Subjects with disease progression at 6 weeks who do not have significant toxicities may remain on therapy for an additional six weeks until a progression is confirmed. Further study drug administration beyond 12 weeks will be at the discretion of the investigator provided that the subject does not have disease progression, does not have unacceptable side effects, does not withdraw from study, or does not have a medical condition or illness that renders the subject unacceptable to receive further study drug.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib is available in capsule form. The dose is 60 mg daily by mouth. Subjects with disease progression at 6 weeks who do not have significant toxicities may remain on therapy for an additional six weeks until a progression is confirmed. Further study drug administration beyond 12 weeks will be at the discretion of the investigator provided that the subject does not have disease progression, does not have unacceptable side effects, does not withdraw from study, or does not have a medical condition or illness that renders the subject unacceptable to receive further study drug.
  Other Names: XL184

SUMMARY:
The purpose of this study is to look at the effects of cabozantinib on castrate-resistant prostate cancer metastatic (cancer that has spread to other parts of the body) to the bone and to learn about any side effects caused by taking cabozantinib.

DETAILED DESCRIPTION:
A significant proportion of patients with prostate cancer develop metastatic disease, which most commonly affects the skeleton. Bone metastases are the cause of significant morbidity and mortality in these patients, and require long-term management. Study participants in this research study will have a diagnosis of castration-resistant prostate cancer metastatic to bone.

Cabozantinib is not approved by the United States Food and Drug Administration (FDA) to treat people for castration-resistant prostate cancer metastatic to bone or for any other type of cancer. Giving cabozantinib to human cancer patients is experimental. Cabozantinib is currently being given to patients on other studies. Cabozantinib is known to have anti-tumor effects and to reduce bone metastases based on early clinical studies in prostate cancer and other cancers. The drug is known to have side effects. The most common side effects were fatigue, diarrhea, anorexia, rash, and palmar-plantar erythrodysesthesia (PPE) syndrome. To date, it is not known if cabozantinib is safe and/or effective.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically and radiologically confirmed castrate-resistant prostate cancer metastatic to bone
* Bone metastases which are accessible for biopsy under CT guidance.
* Willingness to undergo sequential biopsy of bone lesions.
* No prior standard chemotherapy for metastatic disease (neoadjuvant, adjuvant and hormonal treatments are excluded).
* Participant must have discontinued antiandrogen therapy at least 4 weeks (for flutamide and megestrol acetate) or 6 weeks (for bicalutamide or nilutamide) prior to the first dose of XL184. Participants currently on LHRH or GnRH agonists can be maintained on these agents.
* Greater than or equal to 18 years old on day of consent
* Participants must be able to care for themselves
* Adequate organ and bone marrow function
* Participants must be capable of understanding and complying with the protocol requirements and has signed the informed consent document.
* Men capable of sexual activity will be required to agree to use a condom during sexual contact with women having the potential to bear children during their participation in the study and for six months after participation.

Exclusion Criteria:

* Prior therapy with cabozantinib
* Any other type of investigational agent within 28 days before the first dose of study treatment or 5 half-lives of the compound or active metabolite, whichever is longer
* No radiation therapy within 14 days of study treatment. No radionuclide treatment within two months.
* No known brain metastases.
* Test results that measure how quickly blood clots need to be adequate for the study
* Participants who require concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel). Low dose aspirin (≤ 81 mg/day), low-dose warfarin (≤ 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted.
* Participants must not have uncontrolled significant illness including but not limited to: ongoing or active infection requiring systemic treatment, symptomatic congestive heart failure, uncontrolled hypertension , history of hypertensive emergency (e.g.encephalopathy) or hypertensive urgency within 6 months of study treatment, clinically significant wounds including osteonecrosis, history of organ transplant, unstable angina pectoris, stroke within 3 months of study drug, heart attack within 3 months of study drug, development of clots within blood vessels within 6 months of study drug, bleeding from distended veins within 3 months of study drug, any other severe or life threatening hemorrhage/bleeding, major surgery within 4 weeks of study treatment, clinically significant cardiac arrhythmias, history of bowel obstruction within 6 months of study drug or unresolved malabsorption syndrome, untreated bone fracture including tumor-related pathologic fracture, anticipated need for major surgery during the period of the study.
* Corrected QT interval, as measured by an ECG, must be within acceptable protocol limits within 28 days of entering the study
* Unable to swallow capsules
* Unable to undergo MRI
* History of another malignant disease within two years with the exception of superficial skin or bladder cancer which has been completely resected or carcinoma in situ without evidence of invasion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Smith, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabozantinib (XL184)
Started | 25
Completed | 22
Not Completed | 3
Not completed — 25 patients enrolled, 3 were not treated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 67 [56 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Remain Progression-free at 12 Weeks
Description: Efficacy will be measured by the proportion of participants who remain progression-free at 12 weeks after initiation of the study. RECIST 1.1 will be used to measure progression. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, or the appearance of one or more new lesions. Kaplan-Meier methods will be used to report progression-free survival.
Time Frame: 12 weeks after participant initiates study
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 22
Percentage of participants | 77.3 [54.6 to 92.2]

2. Secondary Outcome: Incidence of Adverse Events (AEs) Related to Treatment
Description: The incidence of grades 1-3 AEs, by CTCAE 4.0 category, either possibly, probably or definitely related to treatment. The NCI Common Terminology Criteria for Adverse Events (CTCAE) is a descriptive terminology which can be utilized for AE reporting.
Time Frame: 18 months
Measure: Number; unit: adverse events reported
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 22
adverse events reported
  Blood and Lymphatic System | 10
  Cardiac | 2
  Ear and Labyrinth | 2
  Endocrine | 4
  Eye | 1
  Gastrointestinal | 68
  General and Administrative Site Conditions | 18
  Immune System | 1
  Infections | 7
  Injury | 2
  Investigations | 78
  Metabolism and Nutrition | 29
  Musculoskeletal and Soft Tissue | 8
  Nervous System | 19
  Psychiatric | 2
  Renal and Urinary | 12
  Reproductive and Breast | 1
  Respiratory, Thoracic and Mediastinal | 17
  Skin and Subcutaneous | 24
  Vascular | 11

3. Secondary Outcome: Mean Fold Change in Bone Metabolism Biomarker Expression With Cabozantinib
Description: Mean fold change in markers of bone metabolism in bone and serum with cabozantinib. Bone biomarkers include Osteocalcin, NTx, TRAcP, BMP2, SOST, BAP, CICP
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 22
unitless
  Osteocalcin | -3.3 (5.8)
  NTx | 0.5 (15.4)
  TRAcP | -0.1 (2.4)
  BMP2 | 65.5 (49.1)
  SOST | -29.8 (94.5)
  BAP | -1.36 (56.6)
  CICP | 4.8 (80.6)

4. Secondary Outcome: Progression-free Survival
Description: The percentage of participants alive without progression at 12 weeks
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 22
percentage of participants | 89.5 [64.1 to 97.3]

5. Secondary Outcome: Response Proportion in Both Soft Tissue and Bone Disease.
Description: The percentage of participants that respond in soft tissue and bone disease.
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 22
percentage of participants
  Soft Tissue | 5
  Bone Disease | 59

6. Secondary Outcome: Duration of Response.
Description: Duration of response in soft tissue and bone.
Time Frame: 18 months
Measure: Median (Full Range); unit: weeks
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 22
weeks
  Soft Tissue (only one responder) | 9 [9 to 9]
  Bone | 18 [6 to 80]

7. Secondary Outcome: The Number of Patients That Are Progression Free by PSA
Description: The number of patients that are progression free by PSA at 12 weeks
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 22
Participants | 8

8. Secondary Outcome: Median Time to PSA Progression
Time Frame: 18 months
Measure: Median (Full Range); unit: weeks
Arm/Group | Cabozantinib (XL184)
Number analyzed (Participants) | 22
weeks | 6 [6 to 84]

ADVERSE EVENTS:
Arm/Group | Cabozantinib (XL184)
Serious Adverse Events (participants affected / at risk) | 16/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (XL184) (N=22)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) — Cardiac disorders not specifically known
Myocardial infarction (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myelitis (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) — Nervous system disorders not specifically known
Somnolence (Nervous system disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (XL184) (N=22)
Anemia (Blood and lymphatic system disorders) | 11 (15)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 3 (3)
Blurred vision (Eye disorders) | 2 (2)
Cataract (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Anal mucositis (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (12)
Diarrhea (Gastrointestinal disorders) | 16 (32)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Gastrointestinal disorders not specifically known
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (11)
Oral dysesthesia (Gastrointestinal disorders) | 6 (6)
Oral pain (Gastrointestinal disorders) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 12 (19)
Fever (General disorders) | 3 (3)
Flu like symptoms (General disorders) | 1 (2)
Localized edema (General disorders) | 1 (3)
Non-cardiac chest pain (General disorders) | 3 (3)
Pain (General disorders) | 7 (10)
Serum sickness (Immune system disorders) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Penile infection (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (4)
Bruising (Injury, poisoning and procedural complications) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 15 (28)
Alkaline phosphatase increased (Investigations) | 7 (14)
Aspartate aminotransferase increased (Investigations) | 15 (29)
Blood bilirubin increased (Investigations) | 2 (5)
Creatinine increased (Investigations) | 2 (2)
Investigations - Other, specify (Investigations) | 4 (4)
Lipase increased (Investigations) | 7 (12)
Lymphocyte count decreased (Investigations) | 5 (6)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 7 (7)
Serum amylase increased (Investigations) | 3 (3)
Weight loss (Investigations) | 11 (15)
White blood cell decreased (Investigations) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 17 (23)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Musculoskeletal and connective tissue disorders not specifically known
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7)
Concentration impairment (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (6)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 13 (18)
Headache (Nervous system disorders) | 3 (3)
Myelitis (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) — Psychiatric disorders not specifically known
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 6 (6)
Proteinuria (Renal and urinary disorders) | 7 (8)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (3) — Renal and urinary disorders not specifically known
Renal calculi (Renal and urinary disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Skin and subcutaneous tissue disorders not specifically known
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 4 (6)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 4 (5)
Hypertension (Vascular disorders) | 5 (7)
Vascular disorders - Other (Vascular disorders) | 1 (1) — Vascular disorders not specifically known

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes